CLINICAL TRIAL: NCT06083753
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Multicenter Study to Evaluate the Safety and Efficacy of Oral PIPE-307 as an Adjunctive Treatment in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Study to Evaluate the Safety and Efficacy of PIPE-307 in Subjects With Relapsing-Remitting Multiple Sclerosis
Acronym: VISTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PIPE 307-201
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; PIPE 307; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PIPE-307 Dose A (Experimental)
  Interventions: Drug: PIPE-307 Dose A
- PIPE-307 Dose B (Experimental)
  Interventions: Drug: PIPE-307 Dose B
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PIPE-307 Dose A — Subjects will receive daily oral doses of PIPE-307
  Arms: PIPE-307 Dose A
Drug: PIPE-307 Dose B — Subjects will receive daily oral doses of PIPE-307
  Arms: PIPE-307 Dose B
Drug: Placebo — Subjects will receive daily oral matching dose of Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind study of PIPE-307 or placebo in subjects with relapsing-remitting multiple sclerosis. Subjects will be randomized into 1 of 3 separate cohorts (1:1:1 randomization ratio, PIPE-307 Dose A:PIPE-307 Dose B: Placebo) for a total duration of approximately 30 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind study of PIPE-307 or placebo given to 168 subjects randomized into one of 3 separate cohorts. They will be randomized 1:1:1 (PIPE-307 Dose A:Pipe 307 Dose B: Placebo). There will be a 28-day screening period followed by a 26-week treatment period. Safety will be assessed by periodic measurements of vital signs (VS), physical (PE) and neurological examinations, electrocardiograms (ECG), blood laboratory analyses and occurrence of adverse events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subject is fluent in English.
* Male or female 18 to 50 years of age, inclusive, at the first Screening visit.
* A diagnosis of relapsing-remitting multiple sclerosis (RRMS) according to the 2017 Revised McDonald Criteria.
* Expanded Disability Status Scale (EDSS) and retinal nerve fiber layer within protocol requirements.
* Stable immunomodulatory treatment on no more than a single DMT for RRMS over the 6 months prior to Screening, as determined by the PI.
* Male or female subjects with reproductive potential agree to comply with a highly effective contraceptive method as per protocol through 1 month after last study drug administration as per protocol.
* General good medical health with no clinically significant or relevant abnormalities except those attributed to the underlying multiple sclerosis (MS), including medical history, physical exam, vital signs, ECG and laboratory evaluations, as assessed by the Investigator.

If enrolled in the visual evoked potential (VEP) sub-study, an additional inclusion criterion includes:

- Screening VEP P100 latency greater than the upper limit of normal (as defined in the protocol) in at least one eye, OR a protocol-defined difference in VEP P100 latency between eyes.

Exclusion Criteria:

* Diagnosis or history of symptoms of optic neuritis within 9 months prior to Screening in either eye.
* Diagnosis of MS more than 10 years prior to Screening.
* History of severe myopia, ophthalmologic or retinal disorder that would interfere with measurements of low contrast letter acuity (LCLA) or exam by optical coherence tomography (OCT), as determined by Investigator.
* Concurrent use of dalfampridine or other 4-aminopyridine or diamino-4-aminopyridine drugs.
* Clinical MS relapse or MS related treatment with corticosteroids within 6 months prior to or during Screening.
* History of treatment with bone marrow transplantation, mitoxantrone, cyclophosphamide, atacicept, or irradiation.
* Use of any daily or routine anticholinergic medications within 30 days of Screening or concurrent during the study.
* The presence of gadolinium enhancing lesions by MRI.
* Use of any drugs known to strongly or moderately induce or inhibit Cytochrome P450 3A4 (CYP3A4) enzyme activity within 30 days prior to Screening or concurrent during the study.
* Use of an investigational product, vaccine or intervention other than a non-interventional registry study within the greater of 30 days or 5 half-lives (if known) prior to Screening or expected during the study.
* History of malignancy under current active treatment or considered at substantial risk for progression or recurrence during the study interval, and/or significant cardiac disorder or dysrhythmia, as determined by the Investigator.
* History of a suicide attempt or suicidal behavior or considered at risk for suicide as judged by the PI using the Columbia-Suicide Severity Rating Scale (C-SSRS) as Screening.

If enrolled in the visual evoked potential (VEP) sub-study, an additional exclusion criterion includes:

- History of an ophthalmologic or retinal disorder that would interfere with measurements of VEP, as determined by the Investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAE) | From baseline to week 26 (end of treatment period)
  Number of participants with TEAEs
Change in binocular 2.5% low contrast letter acuity (LCLA) | From baseline to week 26 (end-of-study)

SECONDARY OUTCOMES:
Percentage of subjects with >/=5-letter gain in binocular 2.5% LCLA | From baseline to week 26
Change in monocular 2.5% LCLA | From baseline to week 26
Number of subjects with at least a 15% change in disability with the Timed 25-Foot Walk Test (T25WT) | From baseline to week 26
Number of subjects with at least a 15% change in disability with the Nine-Hole Peg Test (9HPT) | From baseline to week 26
Number of subjects with at least a 15% change in disability with the Symbol Digital Modality Test (SDMT) | From baseline to week 26
Change in magnetic resonance imaging (MRI) measures of myelination and MS disease activity | From baseline to week 26
Change in serum neurofilament light chain (NfL) | From baseline to week 26
Pharmacokinetics: Change in blood concentration levels of PIPE-307 | From baseline to week 30

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — Contineum Therapeutics
Locations (21):
- United States (21):
  - Xenosciences, Phoenix, Arizona
  - Arizona Neuroscience Research, LLC, Phoenix, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - MS and Neuromuscular Center of Excellence, Clearwater, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Shepherd Center, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Neurology Center of New England P.C., Foxborough, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico/Health Science Center/MIND Imaging Center/MS Specialty Clinic, Albuquerque, New Mexico
  - Dent Neurologic Institute, Amherst, New York
  - Neurological Associates of Long Island, P.C., Lake Success, New York
  - Oklahoma Research Foundation - MS Center of Excellence, Oklahoma City, Oklahoma
  - Sibyl Wray Neurology PC, Knoxville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Bhupesh Dihenia, MD, PA, Lubbock, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - UW Medicine MS Center, Seattle, Washington
  - Multicare Neuroscience Center of Washington, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No